CLINICAL TRIAL: NCT03481491
Title: Interactions Between Striatum and Cerebellum in ADCY5 and PRRT2 Dystonias
Acronym: AMEDYST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C16-128; 2017-A01843-50 (Registry Identifier: RCB)
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Dystonia
Keywords: Cerebellum; Striatum; Human; fMRI; Transcranial magnetic stimulation; Genetic dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the TMS procedure (SHAM or real stimulation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham cerebellar stimulation (Sham Comparator): Participants will receive a Sham stimulation (inefficient probe) applied over the cerebellum.
  Interventions: Other: transcranial magnetic stimulation of the cerebellum
- Real cerebellar stimulation (Active Comparator): Participants will receive a real continuous theta burst stimulation (cTBS) applied over the cerebellum.
  Interventions: Other: transcranial magnetic stimulation of the cerebellum

INTERVENTIONS:
Other: transcranial magnetic stimulation of the cerebellum — The intervention will consist in a continuous theta burst stimulation of the cerebellum under neuronavigation.

SUMMARY:
The investigators will study the relationship between the basal ganglia and the cerebellum in dystonia by associating cerebellar stimulations with functional magnetic resonance imaging analysis.

DETAILED DESCRIPTION:
Although dysfunctions in both basal ganglia and cerebellum in dystonia are well documented, the functional relationships between these two important motor control networks remains unclear in the context of dystonia. Here the investigators propose to tackle this issue by associating cerebellar stimulations with functional analysis using fMRI in dystonic patients.

The working hypothesis is that the primary torsion dystonia (PTD) pathophysiology involves dysfunction of striatum that is amplified by dysregulation of the cerebello-thalamo-striatal pathway.

The project is to study dystonia forms resulting primarily from dysfunctions of the striatum (patients with mutation of the ADCY5 gene) and compare them with patients with putative dysfunction of the cerebellum (patients with mutation of the PRRT2 gene) and healthy controls. In these patients, the investigators will look for (1) how cerebello-thalamo striatal pathway can be influenced by striatal dysfunctions and (2) whether cerebellar stimulation may prevent (or worsen?) the disrupted activity in the basal ganglia and (3) whether striatum-related dystonia share the same abnormal network with another form of dystonia resulting from another dysfunction (patients with PRRT2 mutation).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Dystonia
* characterized ADCY5 or PRRT2 mutation
* must have a European Social Security card or a parent having an European Social Security card
* must be older than > 15 years 3 months
* must be able to give informed consent or, for minor patients, parents must be able to give informed consent
* must be able to comply with all study procedures, based on the judgment by the investigator(s).

Exclusion Criteria:

* major depression or any major mental disorders (axis I disorders)
* neurologic disorder other than dystonia
* presence of pacemaker, intracardiac lines, implanted pumps or stimulators, or metal objects inside the eye or skull, cochlear implant
* Permanent makeup of lips or eyelids
* Black large tattoo close to the head
* Severe claustrophobia
* Current pregnancy or breast feeding
* Copper intrauterine device Subjects with one of the following exclusion criteria will not receive cerebellar stimulation
* Open scalp wounds or scalp infection,
* epilepsy or seizures
* Taking at the time of the study: ketamine, antidepressants, ganciclovir, ritonavir, amphetamines, antiemetic.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2024-08-04 (Actual)

PRIMARY OUTCOMES:
Resting state functional connectivity between the cerebellum and the striatum | 6 weeks
  Synchrony between the cerebellum and the striatum, calculated from resting state fMRI done at visit2 will be compared between the 3 groups (healthy controls, ADCY5 patients, PRTT2 patients)

SECONDARY OUTCOMES:
Amplitude of Low Frequency Fluctuation (ALFF) of blood oxygen level-dependent signal in the cerebellum | 6 weeks
  ALFF of Blood oxygen level-dependent signal in the cerebellum will be compared between the 3 groups (healthy controls, ADCY5 patients, PRTT2 patients
Fractional anisotropy (FA) of the cerebello-striatal tract | 1 day
  FA of the disynaptic tract between the cerebellum and the striatum will be compared between the 3 groups.
Creatine concentration in the striatum measured with diffusion weighted spectroscopy. | 6 weeks
  Creatine concentration in the striatum measured from the spectroscopy, will be compared between the 3 groups
Amplitude of Low Frequency Fluctuation (ALFF) of blood oxygen level-dependent signal in the striatum | 6 weeks
  ALFF of Blood oxygen level-dependent signal in the striatum will be compared between the 3 groups (healthy controls, ADCY5 patients, PRTT2 patients
Resting state functional connectivity between the cerebellum and the thalamus | 6 weeks
  Synchrony between the cerebellum and the thalamus, calculated from resting state fMRI done at visit2 will be compared between the 3 groups (healthy controls, ADCY5 patients, PRTT2 patients)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Flamand-Roze, MD, PhD, Principal Investigator — Pitié-Salpêtrière
Locations (1):
- Département de Neurologie, Fédération des Maladies du Système Nerveux, GH Pitié-Salpêtrière, 47 Bd de l'Hôpital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ekmen A, Meneret A, Valabregue R, Beranger B, Worbe Y, Lamy JC, Mehdi S, Herve A, Adanyeguh I, Temiz G, Damier P, Gras D, Roubertie A, Piard J, Navarro V, Mutez E, Riant F, Welniarz Q, Vidailhet M, Lehericy S, Meunier S, Gallea C, Roze E. Cerebellum Dysfunction in Patients With PRRT2-Related Paroxysmal Dyskinesia. Neurology. 2022 Mar 8;98(10):e1077-e1089. doi: 10.1212/WNL.0000000000200060. Epub 2022 Jan 20. PMID 35058336
- [Result] Ekmen A, Doulazmi M, Meneret A, Jegatheesan P, Herve A, Damier P, Gras D, Roubertie A, Piard J, Mutez E, Tarrano C, Welniarz Q, Vidailhet M, Worbe Y, Gallea C, Roze E. Non-Motor Symptoms and Quality of Life in Patients with PRRT2-Related Paroxysmal Kinesigenic Dyskinesia. Mov Disord Clin Pract. 2023 Jun 5;10(7):1082-1089. doi: 10.1002/mdc3.13795. eCollection 2023 Jul. PMID 37476308